CLINICAL TRIAL: NCT06592677
Title: Early Support After Exposure to Trauma
Acronym: EASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: Regional Centre - Violence, Trauma and Suicide Prevention - Region East (RVTS-East) (Unknown); NORCE Norwegian Research Centre AS (Other); Karolinska Institutet (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 302302
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Post-traumatic Stress Disorder
Keywords: CIPE; PTSD; Indicated prevention; Prolonged Exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Parallel two-armed multicenter add on randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator: senior statistician will be blinded for condition. Junior statistician will not, due to practical barriers (double role as the study coordinator). The person responsible for randomization will be blinded for the outcome of the screening (T0) and baseline (T1) assessments.
  Outcome assessors: graduate psychology students who will perform the clinical interviews will be blinded for condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condensed internet-delivered prolonged exposure (CIPE) + Treatment-as-usual (TAU) (Experimental): Participants in this condition will receive Treatment-as-usual (TAU) from psychosocial crisis teams throughout the entire participation period (1 year post trauma), in addition to CIPE as an add-on lasting for six weeks after randomization (T1; randomization from 4 to 7 weeks, dependent on when the participant is recruited). In CIPE, participants are encouraged to have daily contact with their therapist through a secured email system within the platform. Therapists are also available for phone sessions. Total therapist contact for each participant is generally less than 60 minutes during the whole program. Participants are expected to work on intervention tasks for six hours each week and to complete the intervention in three weeks. The intervention is delivered by psychosocial crisis teams' staff in 14 municipalities in the central-eastern part of Norway. Content, frequency, and quantity of the CIPE+TAU-condition will be measured.
  Interventions: Behavioral: Condensed internet-delivered prolonged exposure (CIPE); Behavioral: Treatment-as-usual (TAU)
- Treatment-as-usual (TAU) only (Active Comparator): Participants in this condition will receive Treatment-as-usual (TAU) throughout the entire participation period (1 year post trauma). The TAU-condition is delivered by the same municipality psychosocial crisis teams as the Condensed internet-delivered prolonged exposure (CIPE) +TAU arm. The crisis teams follow a national guideline (The Norwegian Directorate of Health, 2016), recommending proactive contact with victims, screening for psychosocial difficulties, and offering interventions to individuals with significant levels of trauma-related problems. Most municipalities organize interdisciplinary crisis services consisting of physicians, police, priests, nurses, and psychologists who receive referrals from emergency services after a traumatic event. There is currently considerable heterogeneity in the frequenzy and quantity of intervention across municipalities.
  Interventions: Behavioral: Treatment-as-usual (TAU)

INTERVENTIONS:
Behavioral: Condensed internet-delivered prolonged exposure (CIPE) — 'Condensed Internet-delivered Prolonged Exposure' (CIPE) is an intervention designed for victims with symptoms of post-traumatic stress disorder (PTSD) soon after a traumatic incident. CIPE is a therapist-supported intervention that consists of four modules delivered over the internet. Central CIPE-interventions include psychoeducation of normal post-traumatic reactions, in-vivo exposure, imaginary exposure, and a breathing exercise.
  Arms: Condensed internet-delivered prolonged exposure (CIPE) + Treatment-as-usual (TAU)
Behavioral: Treatment-as-usual (TAU) — There is currently considerable heterogeneity regarding the interventional principles applied in the Treatment-as-usual (TAU) condition across municipal crisis teams. The national guidelines (The Norwegian Directorate of Health, 2016), recommends several interventional principles such as psychological first aid (PFA), psychoeducation regarding crisis reactions/symptoms of acute stress, normalization of such reactions, activation of social support, and practical assistance.

SUMMARY:
A significant proportion of people who are exposed to traumatic events suffer from post-traumatic sequelae, such as post-traumatic stress disorder (PTSD). Indicated preventive interventions soon after trauma could be appropriate. Yet, there is limited evidence for the efficacy of such interventions. Moreover, no evidence-based preventive interventions are readily available for victims in the aftermath of crises and disasters in Norway. Condensed Internet-delivered Prolonged Exposure (CIPE) is a preventive intervention designed for victims with symptoms of PTSD (PTSS) approximately one month after a traumatic event. The treatment is an internet-delivered, therapist assisted intervention, based on principles from Prolonged Exposure. CIPE has proven to be feasible, safe, and effective in previous studies. This study aims to test the effectiveness and cost-effectiveness of CIPE in the context of psychosocial crisis services in Norwegian municipalities.

Hypotheses Effectiveness H1 Participants receiving CIPE + treatment as usual (TAU) will have significantly less PTSS than participants receiving TAU at 6 weeks post T1, and at 6-, and 12- months after the traumatic incident.

H2 Significantly fewer participants receiving CIPE+TAU will fulfill the criteria for PTSD compared to participants receiving TAU, at 6- and 12-months post trauma.

H3 Participants receiving CIPE+TAU will have significantly less symptoms of depression and insomnia than participants receiving TAU at 6 weeks post T1, and at 6-, and 12- months after the traumatic incident.

H4 Participants in the CIPE+TAU-condition will report significantly higher treatment satisfaction at post-treatment, compared to those in the TAU-condition.

H5 Participants with traumatic loss receiving CIPE+TAU will have significantly less symptoms of prolonged grief than such participants receiving TAU 12 months after the loss.

Cost-effectiveness H6 Fewer participants in the CIPE+TAU-condition will be referred to second-tier specialty mental health services, and more will achieve improved quality of life within the first year after the traumatic incident, compared to participants in the TAU-condition.

H7 The CIPE+TAU implementation is more cost-effective compared to the TAU in the short run and may even dominate TAU in the long run (i.e., more effective and less costly).

ELIGIBILITY:
Inclusion Criteria:

* Receives support from a municipal crisis team
* Exposure to a traumatic event (as defined by criteria A for the diagnosis of post-traumatic stress disorder (PTSD) in the DSM-5) within the last seven weeks before randomization
* A total score of 10 or above on the PTSD Symptom Checklist-5 at the time of randomization
* Age 16 or above
* Written informed consent
* Writes and speaks English and/or Norwegian

Exclusion Criteria:

* Severe psychopathology in need of specialized health care (e.g., psychotic symptoms, or high suicide risk) or substance dependence syndrome in need of specialized health care
* Known or evident severe cognitive impairment
* Ongoing traumatization, violence, or threats
* Unstable dose of psychotropic medication two weeks prior to randomization
* Concurrent therapy elsewhere before randomization

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5; Norwegian version) | Post-treatment (10 - 13 weeks after trauma)
  20-item questionnaire that measures DSM-5-specified symptoms of post-traumatic stress disorder (PTSD). The total score ranges from 0 to 80, with higher scores indicating more severe symptoms. Items are rated on a 0 ("not at all") to 4 ("extremely") Likert type scale. The PCL-5 has demonstrated satisfactory psychometric properties in various trauma populations. This study will administer a Norwegian version of the PCL-5. Recall period: one month.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5; Norwegian version) | 6 months follow-up
  20-item questionnaire that measures DSM-5-specified symptoms of post-traumatic stress disorder (PTSD). The total score ranges from 0 to 80, with higher scores indicating more severe symptoms. Items are rated on a 0 ("not at all") to 4 ("extremely") Likert type scale. The PCL-5 has demonstrated satisfactory psychometric properties in various trauma populations. This study will administer a Norwegian version of the PCL-5. Recall period: one month.
PTSD Checklist for DSM-5 (PCL-5; Norwegian version) | 12 months follow-up
  20-item questionnaire that measures DSM-5-specified symptoms of post-traumatic stress disorder (PTSD). The total score ranges from 0 to 80, with higher scores indicating more severe symptoms. Items are rated on a 0 ("not at all") to 4 ("extremely") Likert type scale. The PCL-5 has demonstrated satisfactory psychometric properties in various trauma populations. This study will administer a Norwegian version of the PCL-5. Recall period: one month.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Norwegian version) | 6-months follow-up
  30-item structured interview, developed to assess current and life-time post-traumatic stress disorder (PTSD)-diagnosis, as well as past-week PTSD symptoms. The instrument measures the 20 DSM-5 PTSD-symptoms, in addition to the onset and duration of symptoms, related subjective distress and functional impairment (social, occupational), amongst other aspects of the disorder. Standardized questions and probes are provided. A Norwegian version of the CAPS-5 are administered. CAPS-5 has demonstrated excellent psychometric properties.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Norwegian version) | 12-months follow-up
  30-item structured interview, developed to assess current and life-time post-traumatic stress disorder (PTSD)-diagnosis, as well as past-week PTSD symptoms. The instrument measures the 20 DSM-5 PTSD-symptoms, in addition to the onset and duration of symptoms, related subjective distress and functional impairment (social, occupational), amongst other aspects of the disorder. Standardized questions and probes are provided. A Norwegian version of the CAPS-5 are administered. CAPS-5 has demonstrated excellent psychometric properties.
Patient Health Questionnaire (PHQ-9; Norwegian version) | Post-treatment (10 - 13 weeks after trauma)
  9-item self-report measure of depressive symptom severity. The recall period is 2 weeks. Response is given on a 4-point Likert scale (0: not at all, 1: several days, 2: more than half the days, and 3: nearly every day), resulting in the total score ranging from 0 to 27. Higher scores indicate higher symptom severity. The instrument is sensitive for both clinical- and sub-clinical levels of depressive symptoms, and have demonstrated favorable psychometric properties. A validated Norwegian version of the PHQ-9 is applied.
Patient Health Questionnaire (PHQ-9; Norwegian version) | 6-months follow-up
  9-item self-report measure of depressive symptom severity. The recall period is 2 weeks. Response is given on a 4-point Likert scale (0: not at all, 1: several days, 2: more than half the days, and 3: nearly every day), resulting in the total score ranging from 0 to 27. Higher scores indicate higher symptom severity. The instrument is sensitive for both clinical- and sub-clinical levels of depressive symptoms, and have demonstrated favorable psychometric properties. A validated Norwegian version of the PHQ-9 is applied.
Patient Health Questionnaire (PHQ-9; Norwegian version) | 12-months follow-up
  9-item self-report measure of depressive symptom severity. The recall period is 2 weeks. Response is given on a 4-point Likert scale (0: not at all, 1: several days, 2: more than half the days, and 3: nearly every day), resulting in the total score ranging from 0 to 27. Higher scores indicate higher symptom severity. The instrument is sensitive for both clinical- and sub-clinical levels of depressive symptoms, and have demonstrated favorable psychometric properties. A validated Norwegian version of the PHQ-9 is applied.
Insomnia Severity Index (ISI; Norwegian version) | Post-treatment (10 - 13 weeks after trauma)
  7-item questionnaire, which measures insomnia symptoms during the past two weeks. The instrument utilizes a 5-point Likert scale ranging from 0 to 4, yielding a total score of 0-28. Higher scores indicate more insomnia symptoms. The ISI has demonstrated favorable psychometric properties. A Norwegian version of the ISI is applied.
Insomnia Severity Index (ISI; Norwegian version) | 6-months follow-up
  7-item questionnaire, which measures insomnia symptoms during the past two weeks. The instrument utilizes a 5-point Likert scale ranging from 0 to 4, yielding a total score of 0-28. Higher scores indicate more insomnia symptoms. The ISI has demonstrated favorable psychometric properties. A Norwegian version of the ISI is applied.
Insomnia Severity Index (ISI; Norwegian version) | 12-months follow-up
  7-item questionnaire, which measures insomnia symptoms during the past two weeks. The instrument utilizes a 5-point Likert scale ranging from 0 to 4, yielding a total score of 0-28. Higher scores indicate more insomnia symptoms. The ISI has demonstrated favorable psychometric properties. A Norwegian version of the ISI is applied.
Client Satisfaction Questionnaire (CSQ-8; Norwegian version) | Post-treatment (10 - 13 weeks after trauma)
  Eight-item measure of participants' service satisfaction. Response is given on a scale ranging from one to four, with a resulting total score range from eight to 32. Higher scores suggest higher service satisfaction. A validated Norwegian version of the CSQ-8 will be applied.
EQ-5D-5L (Norwegian version) | Post-treatment (10 - 13 weeks after trauma)
  Self-reported health-related quality of life. Self-care, mobility, pain/discomfort, usual activities, and anxiety/depression are measured on a 5-point scale. Response to each item is given by checking off one of five descriptions of functionality in that domain (e.g., have no problems doing my usual activities, slight problems, moderate problems, severe problems, or unable to do my usual activities). The total score ranges from 5 to 25, with higher scores indicating poorer health-related quality of life. Participant also rate their overall health on a scale from 1 (worst health) to 100 (best health). This scale is called the EQ VAS and is a part of the EQ-5D-5L. The instrument has demonstrated excellent psychometric properties. Recall period: today.
EQ-5D-5L (Norwegian version) | 6-months follow-up
  Self-reported health-related quality of life. Self-care, mobility, pain/discomfort, usual activities, and anxiety/depression are measured on a 5-point scale. Response to each item is given by checking off one of five descriptions of functionality in that domain (e.g., have no problems doing my usual activities, slight problems, moderate problems, severe problems, or unable to do my usual activities). The total score ranges from 5 to 25, with higher scores indicating poorer health-related quality of life. Participant also rate their overall health on a scale from 1 (worst health) to 100 (best health). This scale is called the EQ VAS and is a part of the EQ-5D-5L. The instrument has demonstrated excellent psychometric properties. Recall period: today.
EQ-5D-5L (Norwegian version) | 12-months follow-up
  Self-reported health-related quality of life. Self-care, mobility, pain/discomfort, usual activities, and anxiety/depression are measured on a 5-point scale. Response to each item is given by checking off one of five descriptions of functionality in that domain (e.g., have no problems doing my usual activities, slight problems, moderate problems, severe problems, or unable to do my usual activities). The total score ranges from 5 to 25, with higher scores indicating poorer health-related quality of life. Participant also rate their overall health on a scale from 1 (worst health) to 100 (best health). This scale is called the EQ VAS and is a part of the EQ-5D-5L. The instrument has demonstrated excellent psychometric properties. Recall period: today.
The Recovering Quality of Life (ReQoL; Norwegian version) | Post-treatment (10 - 13 weeks after trauma)
  Validated 10-item self-report measure of quality of life specific to people with different mental health conditions. The total score ranges from 0 to 40, with lower scores indicating low quality of life. The scale has demonstrated excellent psychometric properties.
The Recovering Quality of Life (ReQoL; Norwegian version) | 6-months follow-up
  Validated 10-item self-report measure of quality of life specific to people with different mental health conditions. The total score ranges from 0 to 40, with lower scores indicating low quality of life. The scale has demonstrated excellent psychometric properties.
The Recovering Quality of Life (ReQoL; Norwegian version) | 12-months follow-up
  Validated 10-item self-report measure of quality of life specific to people with different mental health conditions. The total score ranges from 0 to 40, with lower scores indicating low quality of life. The scale has demonstrated excellent psychometric properties.
Traumatic grief inventory self report, TGI-SR+ | 12-months follow-up
  The TGI-SR+ is a 22-item self-report questionnaire to assess symptoms of DSM-5 persistent complex bereavement disorder (PCBD), and ICD-11 Prolonged grief disorder (PGD). Total score ranges from 22 to 110, with higher scores indicating more severe symptoms. The instrument has demonstrated good psychometric properties. Recall period: last month.

OTHER OUTCOMES:
Mild-moderate adverse events questionnaire | Post-treatment (10 - 13 weeks after trauma)
  Severe adverse events are monitored and addressed continuously, and will be reported. Mild-moderate adverse events (AE) are reported on an unvalidated generic questionnaire, utilized in previous studies. Participants are asked to report experiences of AEs, and to describe the event briefly, report number of weeks after the traumatic event when the AE took place, frequency, and duration of the AE, and how the AE impacted quality of life when it occurred and today. The participants are also asked to report an appraisal of whether the AE was associated with receiving Condensed internet-delivered prolonged exposure (CIPE). Recall period: last 6 weeks.
Self-reported work absence and use of health services | Post-treatment (10 weeks after trauma)
  Unvalidated questionnaire measuring job status, number of days on sick leave, annually household income, number of consultations with different types of health professionals, number of days admitted to inpatient psychiatric care, and psychotropic medication. Work absence and the type and quantity of services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 6 weeks (except annual income).
Self-reported work absence and use of health services | 6-months follow-up
  Unvalidated questionnaire measuring job status, number of days on sick leave, annually household income, number of consultations with different types of health professionals, number of days admitted to inpatient psychiatric care, and psychotropic medication. Work absence and the type and quantity of services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 3,5 months (except annual income).
Self-reported work absence and use of health services | 12-months follow-up
  Unvalidated questionnaire measuring job status, number of days on sick leave, annually household income, number of consultations with different types of health professionals, number of days admitted to inpatient psychiatric care, and psychotropic medication. Work absence and the type and quantity of services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 6 months (except annual income).
Clinician-reported use of municipality health services | 2-months follow-up (2 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 3-months follow-up (3 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 4-months follow-up (4 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 5-months follow-up (5 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 6-months follow-up (6 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 7-months follow-up (7 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 8-months follow-up (8 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 9-months follow-up (9 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 10-months follow-up (10 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 11-months follow-up (11 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Clinician-reported use of municipality health services | 12-months follow-up (12 months after trauma)
  Unvalidated questionnaire where clinicians in the municipality health services register date and place of consultation, type of health service, the clinician's profession, content, total minutes used, and any referral to other health services. Use of municipality health services will be transformed to reflect costs related to services used, using cost units from the corresponding financial years. Recall period: 1 month.
Registry data on use of specialist health services | 12-months follow-up
  Registry data from the Norwegian Patient Registry (NPR) on referrals to specialist health services, date of consultation, type of consultation, diagnostic information.
Registry data on use of health services | 12-months follow-up
  Registry data from municipality patient' and user registry (KPR) on consultations with general practitioners and acute health services, date of consultation, type of consultation, diagnostic information.
Registry data on use of health service and work absence | 12-months follow-up
  Registry data on work absence/received social security (FD-Trygd).

CONTACTS AND LOCATIONS:
Overall Officials: Harald Bækkelund, PhD, Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies
Locations (21):
- Norway (21):
  - Asker municipality - Psychosocial crisis team, Asker, Asker
  - Norwegian Center for Violence and Traumatic Stress Studies, Oslo, Oslo County
  - Aurskog-Høland - Psychosocial crisis team, Bjørkelangen
  - Fredrikstad municipality - Psychosocial Crisis team, Fredrikstad
  - Gjøvik municipality - psychosocial crisis team, Gjøvik
  - Halden Municipality - psychosocial crisis team, Halden
  - Hamar Municipality - psychosocial crisis team, Hamar
  - Søndre Land municipality - psychosocial crisis team, Hov
  - Ullensaker municipality - psychosocial crisis team, Jessheim
  - Østre Toten municipality - Psychosocial crisis team, Lena
  - Psychosocial crisis team - Oslo, Bjerke, Oslo
  - Psychosocial crisis team - Oslo, Frogner, Oslo
  - Psychosocial crisis team - Oslo, gamle Oslo, Oslo
  - Psychosocial crisis team - Oslo, Grünerløkka, Oslo
  - Psychosocial crisis team - Oslo, Nordstrand, Oslo
  - Psychosocial crisis team - Oslo, Sagene, Oslo
  - Psychosocial crisis team - Oslo, Stovner, Oslo
  - Psychosocial emergency service - Oslo emergency room, Oslo
  - Ringsaker municipality - Psychosocial crisis team, Ringsaker
  - Gjerdrum - psychosocial crisis team, Sørum
  - Nannestad municipality - psychosocial crisis team, Teigebyen

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant outcome- and background data, and code generated from the project, will be made available upon reasonable request, to the degree permitted by ethical board approval.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning six months and ending 5 years following article production.
Access Criteria: Researchers with a methodologically sound proposal. Proposals should be directed to PI.

REFERENCES:
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Mekawi Y, Silverstein MW, Walker A, Ishiekwene M, Carter S, Michopoulos V, Stevens JS, Powers A. Examining the psychometric properties of the PCL-5 in a black community sample using item response theory. J Anxiety Disord. 2022 Apr;87:102555. doi: 10.1016/j.janxdis.2022.102555. Epub 2022 Mar 10. PMID 35338915
- [Background] Sveen J, Bondjers K, Willebrand M. Psychometric properties of the PTSD Checklist for DSM-5: a pilot study. Eur J Psychotraumatol. 2016 Apr 19;7:30165. doi: 10.3402/ejpt.v7.30165. eCollection 2016. PMID 27098450
- [Background] Marx BP, Lee DJ, Norman SB, Bovin MJ, Sloan DM, Weathers FW, Keane TM, Schnurr PP. Reliable and clinically significant change in the clinician-administered PTSD Scale for DSM-5 and PTSD Checklist for DSM-5 among male veterans. Psychol Assess. 2022 Feb;34(2):197-203. doi: 10.1037/pas0001098. Epub 2021 Dec 23. PMID 34941354
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Brattmyr M, Lindberg MS, Solem S, Hjemdal O, Havnen A. Factor structure, measurement invariance, and concurrent validity of the Patient Health Questionnaire-9 and the Generalized Anxiety Disorder scale-7 in a Norwegian psychiatric outpatient sample. BMC Psychiatry. 2022 Jul 11;22(1):461. doi: 10.1186/s12888-022-04101-z. PMID 35818021
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Wisting L, Johnson SU, Bulik CM, Andreassen OA, Ro O, Bang L. Psychometric properties of the Norwegian version of the Patient Health Questionnaire-9 (PHQ-9) in a large female sample of adults with and without eating disorders. BMC Psychiatry. 2021 Jan 5;21(1):6. doi: 10.1186/s12888-020-03013-0. PMID 33402149
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Buysse DJ, Ancoli-Israel S, Edinger JD, Lichstein KL, Morin CM. Recommendations for a standard research assessment of insomnia. Sleep. 2006 Sep;29(9):1155-73. doi: 10.1093/sleep/29.9.1155. PMID 17040003
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Pedersen H, Havnen A, Brattmyr M, Attkisson CC, Lara-Cabrera ML. A digital Norwegian version of the client satisfaction questionnaire 8: factor validity and internal reliability in outpatient mental health care. BMC Psychiatry. 2022 Oct 31;22(1):671. doi: 10.1186/s12888-022-04281-8. PMID 36316661
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Keetharuth AD, Brazier J, Connell J, Bjorner JB, Carlton J, Taylor Buck E, Ricketts T, McKendrick K, Browne J, Croudace T, Barkham M. Recovering Quality of Life (ReQoL): a new generic self-reported outcome measure for use with people experiencing mental health difficulties. Br J Psychiatry. 2018 Jan;212(1):42-49. doi: 10.1192/bjp.2017.10. PMID 29433611
- [Background] Lenferink LIM, Eisma MC, Smid GE, de Keijser J, Boelen PA. Valid measurement of DSM-5 persistent complex bereavement disorder and DSM-5-TR and ICD-11 prolonged grief disorder: The Traumatic Grief Inventory-Self Report Plus (TGI-SR+). Compr Psychiatry. 2022 Jan;112:152281. doi: 10.1016/j.comppsych.2021.152281. Epub 2021 Oct 21. PMID 34700189
- [Background] Bragesjo M, Arnberg FK, Olofsdotter Lauri K, Aspvall K, Sarnholm J, Andersson E. Condensed Internet-delivered prolonged exposure provided soon after trauma: a randomised trial. Psychol Med. 2023 Apr;53(5):1989-1998. doi: 10.1017/S0033291721003706. Epub 2021 Sep 14. PMID 37310324
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). https://doi.org/10.1176/appi.books.9780890425596
- [Derived] Lassen ER, Birkeland MS, Egeland K, Stene LE, Brodersen D, Ekornas B, Reinholdt NP, Kjerstad E, Lamu AN, Aarons GA, Crable EL, Bragesjo M, Baekkelund H. Early Support after Exposure to Trauma (EASE): protocol for a hybrid effectiveness-implementation trial of an internet-based intervention for PTSD prevention. Trials. 2026 Feb 5. doi: 10.1186/s13063-026-09502-z. Online ahead of print. PMID 41645255
- See also: The Norwegian Directorate of Health. (2016). National guidelines for psychosocial support in the aftermath of crises and catastrophes — https://www.helsedirektoratet.no/veiledere/psykososiale-tiltak-ved-kriser-ulykker-og-katastrofer
- See also: Heir, T. (2014). PCL-5. Norwegian centre for violence and traumatic stress studies. — https://www.nkvts.no//content/uploads/2022/11/Traume-og-PTSD-screening-TRAPS-I.pdf
- See also: Bækkelund, H., Aareskjold, J., & Endsjø, M. (2015). KLINIKERADMINISTRERT PTSD-SKALA FOR DSM-5: Versjon for vurdering av siste måned. Norwegian Centre for Violence and Traumatic Stress Studies. — https://www.nkvts.no//content/uploads/2018/03/KLINIKERADMINISTRERT-PTSD-SKALA-FOR-DSM-5-KAPS-5.pdf